CLINICAL TRIAL: NCT04906889
Title: The Effect of Opioid-free Anesthesia Using Dexmedetomidine-lidocaine on Acute Postoperative Pain in Gynecological Laparoscopy
Brief Title: the Effect of Dexmedetomidine and Licodaine on Acute Postoperative Pain in Gynecological Laparoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: financial protocol
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: dexmedetomidine-lidocaine
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female | interventions — Dexmedetomidine; Remifentanil; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine-lidocaine (Experimental): The study group receives the dexmedetomidine and lidocaine infusion with general anesthesia for gynecological laparoscopy.
  Interventions: Drug: Dexmedetomidine Hydrochloride; Drug: Lidocaine Hydrochloride
- remifentanil (Active Comparator): The control group receives the remifentanil infusion with general anesthesia for gynecological laparoscopy
  Interventions: Drug: Remifentanil Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — dexmedetomidine iv bolus for 10 minutes followed by the infusion of 0.1-1 ug/kg/h during general anesthesia
  Other Names: precedex
  Arms: dexmedetomidine-lidocaine
Drug: Remifentanil Hydrochloride — remifentanil iv infusion of 0.5-5 ng/ml (effect site concentration using TCI) during general anesthesia
  Other Names: remifentanil
  Arms: remifentanil
Drug: Lidocaine Hydrochloride — lidocaine iv bolus followed by the infusion of 1.5mg/kg/h during general anesthesia
  Other Names: lidocaine
  Arms: dexmedetomidine-lidocaine

SUMMARY:
The aim of this study is to investigate the effect of opioid-free anesthesia using dexmedetomidine and lidocaine instead of remifentanil infusion, on the acute postoperative pain after the gynecological laparoscopy

DETAILED DESCRIPTION:
This study is performed to investigate the effect of dexmedetomidine and lidocaine the postopeative pain, shivering, nausea and vomiting after the gynecological laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective gynecological laparoscopy

Exclusion Criteria:

* emergent surgery
* cancer surgery
* chronic pain requiring pain killers
* psychiatric disease
* preoperative bradycardia (HR < 50 bpm)
* allergies
* pregnancy or breast feeding

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain in recovery room | 30 minuetes after the completion of surgery
  The pain level is assessed by using NRS (numeric rating scale; 0=no pain , 10=the worst pain)

SECONDARY OUTCOMES:
shivering in recovery room | 30 minuetes after the completion of surgery
  The incidence of shivering is assessed by questioning Yes or No.
postoperative nausea and vomiting (PONV) | 30 minutes after the completion of surgery
  The incidence of PONV is assessed by questioning Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Young Eun Moon, MD, PhD, Principal Investigator — Associate professor, Department of Anesthesiology and Pain Medicine
Locations (2):
- South Korea (2):
  - Seoul St.Mary's Hospital, Seoul, Seocho-gu
  - Seoul St.Mary's Hospital, Seocho

IPD SHARING:
Plan to Share IPD: No